CLINICAL TRIAL: NCT04132258
Title: "Clinical and Epidemiological Characteristics of Inflammatory Rhinitis in Patients on Biotherapies"
Acronym: RIB18
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC18_0397
Record Dates: First submitted 2019-10-14; First posted 2019-10-18 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Inflammatory Rhinitis
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: survey — (presence of certain antecedents, weight, height, current or past existence of inflammatory rhinitis) and a second by the specialist doctor (pathology at the origin of the start of biotherapy, year of beginning of treatment, previous biotherapies over the last 3 years).

SUMMARY:
Inflammatory rhinitis is a side effect observed in patients treated with biotherapies in the context of chronic bowel disease (IBD) or spondylartrhopathy (SPA). This damage is still poorly described in the literature. I The objective of this study is to study the associated characteristics of crustal rhinitis in a cohort of patients treated with biotherapy for chronic inflammatory disease (IBD, SPA, psoriasis).

DETAILED DESCRIPTION:
Inflammatory rhinitis is a side effect observed in patients treated with biotherapies in the context of chronic bowel disease (IBD) or spondylartrhopathy (SPA). This damage is still poorly described in the literature. It can occur in isolation or in association with a fold pustulose table, which differs from the classic fold pustulose described by Cribier et al in autoimmune diseases by the presence of staphylococcus aureus in the pustules. Some authors also describe associated paradoxical psoriasiform reactions or an impetigo. In our experience, this condition is more frequently found in patients treated for IBD or SPA and has a clinically characteristic fissure appearance. Thus, the semiology but also the epidemiology of this crusty rhinitis is still poorly described.

The objective of this study is to study the associated characteristics of crustal rhinitis in a cohort of patients treated with biotherapy for chronic inflammatory disease (IBD, SPA, psoriasis).

Patient recruitment will take place over a one-year period, in a multi-centre manner (Angers and Nantes University Hospital) with prospective data collection in the form of a questionnaire and clinical evaluation during a dermatology consultation planned in the traditional care pathway for the follow-up of patients with skin manifestations during biotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (> 18 years of age),
* Biotherapy treatment: anti TNF, ustekinumab, secukinumab, ixekizumab, Rituximab, vedolizumab, abatacept, inhibitor jak kinase, anti Il1, Anti Il6,
* Biotherapy treatment > 3 months,
* Chronic inflammatory disease: psoriasis, ankylosing spondylitis (SPA), rheumatoid arthritis (RA), Crohn's disease (CD), bleeding rectocolitis (HRC)
* No opposition to the study

Exclusion Criteria:

* Patient under legal protection measure,
* Refusal of the subject to participate in the study,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruitment of patients on biotherapies that meet the inclusion criteria as exhaustively as possible.
  * Major patients, followed at the University Hospital of Angers and Nantes, in the dermatology, gastroenterology and rheumatology departments for chronic inflammatory diseases requiring treatment with biotherapy started at least 3 months ago.
  * Recruitment during consultations in the specialties concerned or in the day hospitals planned for the administration of treatments.
  Translated with www.DeepL.com/Translator
Sampling Method: Non-Probability Sample
Enrollment: 356 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2020-06-19 (Actual); Study Completion 2020-06-19 (Actual)

PRIMARY OUTCOMES:
Prevalence of inflammatory rhinitis | through study completion, an average of 1 year
  Presence of inflammatory rhinitis yes/no

SECONDARY OUTCOMES:
Characteristics associated with Patient-related characteristics in inflammatory rhinitis. | through study completion, an average of 1 year
  * Age
  * Tobacco use yes/no
  * Diabetes yes/no
  * Verneuil disease yes/no
  * Psoriasis yes/no
  * Eczema in childhood yes/no
  * Underlying pathology (type, start year)
  * Previous biotherapies and duration of exposure over the last 3 years yes/no
Characteristics of rhinitis. | through study completion, an average of 1 year
  * Delays between the start of treatment and the onset of symptoms
  * Treatment under which rhinitis occurred
  * Rhinitis stage
  * Permanent or recurring, unilateral or bilateral
  * Associated functional signs (rhinorrhea, pain...)
  * Quality of Life (DLQI)
  * Presence of documented endonasal staphylococcus yes/no
  * Positivity of anti-nuclear antibodies yes/no
  * Type of treatment carried out

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Nantes, France